CLINICAL TRIAL: NCT07252843
Title: Lymphedema Prediction Model in Breast Cancer After Axillary Lymph Node Dissection: A Study of Clinicopathological Factors, Receptor Expression (VEGFR3, TGFBR2), and Genetic Predisposition (GJA4, MET, GATA2)
Brief Title: Integrating Clinical, Protein Expression, and Genetic Markers to Predict Lymphedema in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rizky Ifandriani Putri, MD, Dharmais National Cancer Center Hospital
Other Study IDs: 308/KEPK/IX/2023
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema Arm
Keywords: breast cancer; lymphedema; prediction model
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA from blood samples FFPE of lymphatic tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational ambidirectional cohort study is to develop a prediction model to identify the risk of lymphedema after axillary lymph node dissection (ALND) in patients with breast cancer. The main questions it aims to answer are:

* Can clinicopathological factors predict the development of lymphedema?
* Do protein expression profiles and genetic mutations increase susceptibility to lymphedema?

Participants will:

* Undergo clinical evaluation and indocyanine green (ICG) lymphography to diagnose lymphedema.
* Provide lymphatic tissue and blood samples during ALND surgery for immunohistochemical protein analysis and gene mutation assessment.
* Be followed over time to monitor the onset and progression of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histopathologically confirmed breast cancer
* Undergoing axillary lymph node dissection (ALND)
* Able to undergo indocyanine green (ICG) lymphography examination

Exclusion Criteria:

* Clinical signs of lymphedema prior to surgery, confirmed by clinical assessment and/or ICG lymphography
* History of iodine allergy, asthma, impaired renal function, pregnancy, or breastfeeding
* Incomplete clinical or laboratory data required for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with breast cancer who are undergoing axillary lymph node dissection (ALND) as part of their standard surgical management. Eligible participants are recruited from Dharmais Cancer Hospital and Bogor City Regional General Hospital in Indonesia. Only patients without pre-existing lymphedema and who are able to undergo indocyanine green (ICG) lymphography are enrolled. Both early- and locally advanced breast cancer cases are included, provided clinical data and follow-up assessments can be completed.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of Arm Lymphedema | Up to 24 months post-axillary lymph node dissection
  Development of lymphedema identified through clinical signs and symptoms, confirmed using indocyanine green (ICG) lymphography. The presence or absence of lymphedema will be recorded during follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Rizky Ifandriani Putri, MD, Principal Investigator — Anatomical Pathology Department, Dharmais Cancer Hospital - National Cancer Center
Locations (1):
- Dharmais Cancer Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The datasets analyzed during the current study are available from the corresponding author upon reasonable request.